CLINICAL TRIAL: NCT06823882
Title: The Impact of Floor-rise Training on Fear of Falling and Independent Floor-rise Ability in Older Adults Living in the Community: A Pilot Cluster Randomised Controlled Trial With Multiple Methods.
Brief Title: Practicing Getting Up From the Floor to Reduce Fear of Falling and Improve Floor-Rise Ability in Community-Dwelling Older Adults: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Principal Investigator, Shane Seeley, Doctor of Physiotherapy (DPT) Student, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHP/A23/004
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Fear of Falling; Floor-Rise Ability; Falls; Post-Fall Recovery; Older Adults (65 Years and Older)

STUDY DESIGN:
Intervention Model Description: Cluster Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Floor-Rise Training Group (Experimental): Participants practiced getting up from the floor using a structured approach called the Backward Chaining Method (BCM). Sessions lasted 20 minutes weekly for 5 weeks, led by an instructor.
  Interventions: Behavioral: Floor-Rise Training
- Video Demonstration Group (Active Comparator): Participants watched a 20-minute instructional video called "Upwards and Onwards", available on the NHS Inform website. The video explains how to get up from the floor safely and how to practice. It was divided into shorter sections over 5 weeks, with group discussions ensuring a total of 20 minutes per week.
  Interventions: Behavioral: Video Demonstration

INTERVENTIONS:
Behavioral: Floor-Rise Training — Practicing getting up from the floor using the Backward Chaining Method (BCM) for 20 minutes per week for 5 weeks
  Other Names: Backward Chaining Method
  Arms: Floor-Rise Training Group
Behavioral: Video Demonstration — Watching a 20-min video on floor-rise technique and over 5 weeks, with discussions. This video explains how to get up safely from the floor and how to practice.
  Arms: Video Demonstration Group

SUMMARY:
Goal:

This pilot study aims to determine whether practicing getting down to and standing up from the floor reduces fear of falling (FoF) and improves older adults' ability to complete this task. The study compares this to a control group that watches educational videos on the same topic. This practice is referred to as Floor-Rise Training (FRT).

Main Questions:

1. Can a short FRT intervention reduce fear of falling?
2. Can a short FRT intervention improve the ability to rise from kneeling, sitting, and lying positions?
3. Does watching an instructional video on FRT improve fear of falling or floor-rise ability?

Study Design:

Researchers will compare:

* A group receiving 20 minutes of FRT weekly for 5 weeks.
* A control group watching FRT videos followed by discussions over the same period. Changes in floor-rise ability and FoF will be assessed to determine the effectiveness of FRT.

Participants:

Participants will be recruited from five Otago exercise classes (a falls prevention program without FRT) in Renfrewshire. Each class will be randomly assigned to either:

* The FRT intervention group (3 classes).
* The control group (2 classes) watching videos that include an FRT demonstration. Participants will complete questionnaires (to assess FoF) and timed floor-rise tests before and after the intervention. Some may also be invited to focus groups to share their experiences with the intervention, videos and with our recruitment procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* Able to provide written informed consent
* Currently engaged with ROAR and attending the Otago exercise classes

Exclusion Criteria:

* Requiring a walking frame indoors to mobilise
* Have any medical condition that renders it inadvisable to descend to the floor (e.g. such as awaiting knee replacement surgery)
* Any uncontrolled medical condition requiring medical input
* BM I≥ 30 kg/m2
* Lacking capacity to consent to participate
* Unable to comprehend FRT instructions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Falls Efficacy Scale-International (FES-I) | Baseline and 1 week following the intervention (6 weeks post-baseline).
  A 16-item questionnaire that assesses concern about falling during daily activities. Scores range from 16 (no concern) to 64 (severe concern). A lower score indicates a lower fear of falling.

SECONDARY OUTCOMES:
Timed Floor-Rise (Supine to Standing) | Baseline and 1 week following the intervention (6 weeks post-baseline).
  Time taken (in seconds) for a participant to rise independently from a supine position (lying on their back) to a standing position using a sturdy chair. Faster time indicates improved ability.
Timed Floor-Rise (Sitting to Standing) | Baseline and 1 week following the intervention (6 weeks post-baseline).
  Time taken (in seconds) for a participant to rise from a sitting position on the floor to standing using a sturdy chair. Faster time indicates improved ability.
Timed Floor-Rise (Kneeling to Standing) | Baseline and 1 week following the intervention (6 weeks post-baseline).
  Time taken (in seconds) for a participant to rise from a kneeling position to standing using a sturdy chair. Faster time indicates improved ability.
Perceived Ability to Manage Falls (PAMF) | Baseline and 1 week following the intervention (6 weeks post-baseline).
  The PAMF is a 5-item questionnaire measuring confidence in independently recovering from a fall. Scores range from 4 to 20, with higher scores indicating greater confidence.
Fear of Falling Visual Analog Scale (VAS) - Indoor | Baseline and 1 week following the intervention (6 weeks post-baseline).
  Participants mark with an "x" on a 0-100 scale measuring fear of falling indoors, with higher scores indicating greater fear.
Fear of Falling Visual Analog Scale (VAS) - Outdoor | Baseline and 1 week following the intervention (6 weeks post-baseline).
  Participants mark with an "x" on a 0-100 scale measuring fear of falling outdoors, with higher scores indicating greater fear.
Activity Avoidance (VAS) | Baseline and 1 week following the intervention (6 weeks post-baseline).
  Participants mark with an "x" on a 0-100 scale measuring the percentage of activities avoided due to fear of falling, with higher scores indicating greater avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn A Skelton, PhD, Study Director — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data for primary and secondary outcome measures
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication and ending 5 years after publication.
Access Criteria: Qualified researchers affiliated with academic institutions will be able to access the de-identified participant-level data for primary and secondary outcome measures and study protocol by contacting the principal investigator.